CLINICAL TRIAL: NCT06810895
Title: Evaluation of AK104 (Cadonilimab) Combined with Chemotherapy for Recurrent or Metastatic Small Cell Neuroendocrine Carcinoma of the Cervix: a Single-Arm, Open-Label, Multicenter Clinical Study
Brief Title: Evaluation of AK104 (Cadonilimab) Combined with Chemotherapy for Recurrent or Metastatic Small Cell Neuroendocrine Carcinoma of the Cervix
Status: Enrolling by invitation | Type: Observational
Sponsor: Ding Ma (Other)
Responsible Party: Sponsor-Investigator, Ding Ma, Chairman of Obstetrics & Gynecology department of Tongji hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ22-GYN/SCNEC -01
Record Dates: First submitted 2024-10-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Cervix Cancer; Cadonilimab; Small Cell Neuroendocrine Carcinoma of the Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples, Tissue Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cadonilimab Plus Chemotherapy Group: Participants in this group will receive AK104 (Cadonilimab) combined with chemotherapy (cisplatin or carboplatin, and etoposide) for six cycles. After the chemotherapy phase, participants will continue with AK104 monotherapy until disease progression, intolerable toxicity, or other protocol-defined reasons, for a maximum treatment duration of 24 months.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of AK104 (Cadonilimab) combined with chemotherapy (cisplatin or carboplatin, and etoposide) for the treatment of recurrent or metastatic small cell neuroendocrine carcinoma of the cervix. The main questions it aims to answer are:

Is AK104 (Cadonilimab) combined with chemotherapy effective in treating recurrent or metastatic small cell neuroendocrine carcinoma of the cervix? What side effects or medical issues do participants experience while taking AK104?

Participants will:

Receive AK104 (10 mg/kg) combined with either cisplatin (75 mg/m²) or carboplatin (AUC 5) and etoposide (100 mg/m²) every three weeks for up to six cycles.

After chemotherapy, continue with AK104 (10 mg/kg every three weeks) until disease progression, intolerable toxicity, investigator decision, withdrawal of consent, death, or other reasons specified in the protocol, with a maximum treatment duration of 24 months.

Undergo tumor assessments every 6 weeks (±7 days) for the first 48 weeks after the first dose, and every 12 weeks (±7 days) thereafter.

Participants who discontinue treatment for reasons other than disease progression will continue with follow-up for disease status as much as possible, until they begin another anticancer therapy, experience disease progression, withdraw consent, die, or the study ends, whichever occurs first.

Researchers will evaluate the safety of AK104 by assessing adverse events (AEs) using the NCI CTCAE version 5.0 grading system, and determine their relationship to the drug. Depending on the severity of the AEs and their relationship to the drug, researchers will take appropriate measures and provide additional treatments to ensure participant safety.

After completing treatment, participants will have a safety follow-up visit (90 days after the last dose) and then participate in survival follow-up every 3 months to collect survival information and information on subsequent anticancer treatments until death, withdrawal of consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written Informed Consent Form (ICF).
2. Female participants aged ≥18 years and ≤75 years at the time of enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
4. Histologically or cytologically confirmed small cell neuroendocrine carcinoma of the cervix, classified as recurrent or metastatic, with no prior systemic therapy for the recurrent or metastatic stage. Recurrent patients must be assessed by the investigator as unsuitable for surgery or radiotherapy.
5. At least one untreated measurable lesion according to RECIST v1.1.
6. Adequate organ function:

   a) Hematologic (no use of any blood components or growth factor support within 7 days before starting study treatment): i. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1,500/mm³); ii. Platelet count ≥ 100 × 10^9/L (100,000/mm³); iii. Hemoglobin ≥ 90 g/L. b) Renal: i. Estimated creatinine clearance (CrCl) ≥ 50 mL/min.
   * CrCl will be calculated using the Cockcroft-Gault formula:

   CrCl (mL/min) = {(140 - age) × weight (kg) × 0.85} / (serum creatinine (mg/dL) × 72).

   ii. Urine protein < 2+ or 24-hour urine protein < 1.0 g. c) Hepatic: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN; ii. AST and ALT ≤ 2.5 × ULN; iii. Serum albumin (ALB) ≥ 28 g/L. d) Coagulation: i. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (participants receiving anticoagulation therapy must be on a stable dose, and coagulation parameters (PT/INR and APTT) should be within the expected therapeutic range at screening).

   e) Cardiac function: i. Left ventricular ejection fraction (LVEF) ≥ 50%.
7. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test is required, and the serum result will prevail). If a female participant of childbearing potential is sexually active with a non-sterilized male partner, she must use acceptable contraception starting from screening and agree to continue using contraception for 120 days after the last dose of the study drug; discontinuation of contraception after this point should be discussed with the investigator.
8. Participants must be willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Other pathological histological types (e.g., squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, clear cell carcinoma, sarcoma, etc.).
2. Malignant tumors other than small cell neuroendocrine carcinoma of the cervix within 3 years before enrollment. Participants with other malignancies cured by local treatment, such as basal or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the breast, are not excluded.
3. Concurrent enrollment in another clinical study, unless it is an observational, non-interventional study or the follow-up phase of an interventional study.
4. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment, or autoimmune disease that is likely to recur or require planned treatment as judged by the investigator; exceptions include: skin diseases not requiring systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema); hypothyroidism due to autoimmune thyroiditis requiring only a stable dose of hormone replacement therapy; well-controlled type 1 diabetes mellitus; childhood asthma that has completely resolved without adult intervention; diseases judged by the investigator as unlikely to recur in the absence of external triggers.
5. Active or clinically required treatment of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
6. Requirement for systemic corticosteroids (>10 mg prednisone equivalent per day) or other immunosuppressive drugs within 14 days after taking the study drug. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement doses >10 mg prednisone equivalent per day are allowed. Participants are allowed to use topical, ocular, intra-articular, intranasal, and inhaled corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are allowed even if >10 mg/day of prednisone equivalent. Short-term use of corticosteroids for prevention (e.g., contrast allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions due to contact allergens) is permitted.
7. Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4), immune checkpoint agonists (e.g., antibodies against ICOS, CD40, CD137, GITR, OX40), immune cell therapies, or any treatment targeting tumor immunomodulatory mechanisms.
8. Known history of human immunodeficiency virus (HIV) or positive test for acquired immune deficiency syndrome (AIDS).
9. Known history of allogeneic organ transplant or allogeneic hematopoietic stem cell transplantation.
10. Known history or presence of interstitial lung disease.
11. History of gastrointestinal perforation and/or fistula within 6 months prior to enrollment.
12. Necrotic lesions identified within 4 weeks before enrollment, with a risk of major hemorrhage as judged by the investigator.
13. Severe infection within 4 weeks before the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.
14. Known active tuberculosis (TB). Participants suspected of having active TB should be excluded based on chest X-ray, sputum examination, and clinical symptoms and signs.
15. Untreated chronic hepatitis B or hepatitis B virus (HBV) carriers with HBV DNA >1000 IU/mL, and participants with active hepatitis C should be excluded. Non-active hepatitis B surface antigen (HBsAg) carriers, participants with stable hepatitis B after treatment (HBV DNA <1000 IU/mL), and cured hepatitis C participants can be enrolled. Participants positive for HCV antibodies are eligible only if HCV RNA is negative.
16. Receipt of the last radiotherapy or antitumor therapy (e.g., chemotherapy, targeted therapy, herbal medicine for tumor control, tumor embolization) within 4 weeks before the first dose of AK104.
17. Major surgery within 30 days prior to the first dose of AK104, or failure to recover fully from prior surgery. Local surgery (e.g., placement of a central venous port, core needle biopsy, prostate biopsy) is allowed, provided it is completed at least 24 hours before the first dose of study medication.
18. Known history or presence of meningeal metastasis, spinal cord compression, leptomeningeal disease, or active brain metastases. However, participants who meet the following requirements and have measurable lesions outside the central nervous system may be enrolled: 1) Previously untreated, currently asymptomatic (e.g., no neurological impairment, seizures, or other typical CNS metastasis symptoms and signs; no corticosteroid treatment required); 2) Asymptomatic after treatment with radiographic stability for at least 4 weeks before the start of study treatment (e.g., no new or enlarged brain metastases) and cessation of systemic corticosteroids and antiepileptic therapy for at least 2 weeks.
19. Participants with pleural effusion, pericardial effusion, or ascites that cannot be controlled stably despite repeated drainage or other methods as determined by the investigator.
20. Uncontrolled comorbidities, including symptomatic congestive heart failure (New York Heart Association Classification of Functional Status Class 3 or 4), uncontrolled hypertension, unstable angina, poorly controlled arrhythmias, evidence of acute or active myocardial ischemia, severe active peptic ulcer disease or gastritis, or psychiatric/psychosocial conditions that may limit compliance with study requirements or affect the ability to provide written informed consent. Any arterial thromboembolism, including myocardial infarction, cerebrovascular accident, or transient ischemic attack, within 6 months prior to enrollment, history of deep vein thrombosis, pulmonary embolism, or other serious thromboembolic events.
21. Unresolved toxicity from prior antitumor treatment, defined as toxicity not recovered to Grade 0 or 1 by NCI CTCAE version 5.0, or to the level specified in the inclusion/exclusion criteria, except for alopecia. Participants with irreversible toxicity not expected to be exacerbated by study drug administration (e.g., hearing loss) may be included after consultation with the medical monitor. Participants with irreversible radiation-induced late toxicity may be included after consultation with the medical monitor.
22. Receipt of a live vaccine within 30 days before the first dose of AK104, or planned receipt of a live vaccine during the study.
23. Known history of severe hypersensitivity to other monoclonal antibodies.
24. Known allergy to any components of the AK104 formulation.
25. Pregnant or breastfeeding women.
26. Any condition that, in the opinion of the investigator, may pose a risk to the participant receiving study medication, interfere with the evaluation of study medication, or compromise participant safety or study results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population includes adult female participants aged 18 to 75 years, diagnosed with small cell neuroendocrine carcinoma of the cervix that is recurrent or metastatic. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2 and adequate organ function as defined by laboratory tests. Eligible participants should not have received prior systemic treatment for the recurrent or metastatic stage of the disease. The study excludes participants with other malignancies (unless previously cured by local treatment), active autoimmune diseases requiring systemic therapy, or untreated chronic hepatitis B and C. Participants must be willing to comply with scheduled visits, treatment plans, and laboratory tests throughout the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Cadonilimab Combined with Chemotherapy in Treating Recurrent or Metastatic Small Cell Neuroendocrine Carcinoma of the Cervix | At least 3 months from the start of the study to the end of treatment
  The number of participants who experience treatment-related adverse events (graded according to CTCAE v4.0) during treatment will be measured. Data will include the type, severity, and frequency of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At least 6 months after the end of treatment.
  The percentage of participants achieving either complete response (CR) or partial response (PR), as determined by RECIST v1.1 criteria.
Progression-Free Survival (PFS) | At least 6 months after the end of treatment
  Time from the start of treatment to disease progression or death from any cause, measured using the Kaplan-Meier method. Progression will be determined according to RECIST v1.1 criteria.
Overall Survival (OS) | At least 12 months after the end of treatment.
  Time from the start of treatment to death from any cause, measured using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (1):
- ongji Hospital, Tongji Medical College, Huazhong University of Science andTechnology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes
We will regularly check if new subjects have been recruited into the study and update the data.
Supporting Information: Study Protocol, SAP, ICF, CSR